CLINICAL TRIAL: NCT00004670
Title: Phase II Study of Pallidotomy for Parkinson Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Emory University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/12083; EUSM-018; EUSM-409-92
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Parkinson Disease; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Pallidotomy

INTERVENTIONS:
Procedure: pallidotomy

SUMMARY:
OBJECTIVES:

I. Evaluate the safety and efficacy of pallidotomy immediately following 3 preoperative assessments vs. delayed pallidotomy following 6 months of standard medical therapy in patients with Parkinson disease.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized study. One group of patients undergoes the surgical procedure pallidotomy, a precise lesioning of brain cells in the globus pallidus.

The other group receives standard medical care for 6 months followed by a pallidotomy.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Idiopathic Parkinson disease Hoehn and Yahr stage III or worse during "off" periods

Responsive to levodopa by history or exam Sub-optimal clinical response to maximal medication Medication optimized for at least 4 weeks prior to entry

No atypical or secondary disease, e.g.:

* No history of cerebrovascular accident
* No cerebellar involvement
* No severe brain atrophy on magnetic resonance imaging

No Mattis Dementia Rating Scale score less than 116

No dementia meeting Diagnostic and Statistical Manual of Mental Disorders-IV criteria

No Hamilton Depression Rating Scale score greater than 10

No Hamilton Anxiety Scale score greater than 14

--Patient Characteristics--

Other: No medical contraindication to surgery, e.g.:

* Diabetes
* Cardiopulmonary disease

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 1994-10

CONTACTS AND LOCATIONS:
Overall Officials: Mahlon R. DeLong, Study Chair — Emory University